CLINICAL TRIAL: NCT07299409
Title: A Phase II Study of First-Line Sacituzumab Govitecan in Advanced Untreated Triple-Negative Breast Cancer Patients.
Brief Title: First-Line Sacituzumab Govitecan in Advanced Untreated Triple-Negative Breast Cancer Patients.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nathalie Levasseur (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor-Investigator, Nathalie Levasseur, Medical Oncologist, Principal Investigator, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG6978
Record Dates: First submitted 2025-06-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Triple Negative Breast Cancer; Breast Cancer Metastatic; Breast Cancer
Keywords: advanced breast cancer; Sacituzumab govitecan; genomics; whole-genome and transcriptome analysis; triple negative breast cancer; Personalized OncoGenomics (POG)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Intervention Model Description: This will be a non-randomized phase II single-arm study of first-line Sacituzumab govitecan in participants with advanced triple-negative breast cancer who have not received prior treatment in the advanced setting. Participants will receive an initial dose of SG on Days 1 and 8 of 21-day cycles. Treatment and cycles will continue until there is evidence of disease progression, significant toxicity, or if the participant or Investigator decide to discontinue treatment for any reason.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan (Experimental): Patients will receive SG at an initial dose of 10 mg per kilogram intravenously on day 1 and 8 of 21-day cycles. Treatment and cycles will continue until there is evidence of disease progression, significant toxicity, or if the participant or Investigator decide to discontinue treatment for any reason.
  Interventions: Drug: Sacituzumab Govitecan (SG)

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Administer Sacituzumab Govitecan (SG) at 10 mg/kg as an intravenous (IV) infusion on Days 1 and 8 of a 21-day cycle. SG should not be administered as an IV push or bolus.
  Other Names: Trodelvy

SUMMARY:
The goal of this clinical trial is to learn if the drug Sacituzumab govitecan (SG) reduces disease progression when used as a first-line treatment in adults with advanced triple-negative breast cancer (TNBC) who have not received prior treatments in the advanced setting. It will also look at whether the effectiveness of the drug differs between TNBC adults with homologous recombination deficiency (HRD) subtypes and those with non-HRD subtypes. The main questions this study aims to answer are:

* Will patients with advanced TNBC who haven't received prior treatment in the advanced setting respond better (i.e., slowed disease progression) when given SG as a first-line treatment?
* Does the overall response rate of SG differ between HRD vs non-HRD advanced TNBC patients without prior treatment in the advanced setting?

Participants will:

* Be given drug SG on days 1 and 8 of 21-day cycle(s)
* Will continue (repeat) 21-day cycles until disease progression or voluntary withdrawal
* Visit the clinic for treatments on days 1 and 8
* Have long-term follow-up every 12 weeks via phone or in-clinic

DETAILED DESCRIPTION:
This study is a non-randomized phase II single-arm trial of first-line sacituzumab govitecan (SG) in participants with advanced triple-negative breast cancer who have not received prior treatment in the advanced setting. It is designed to assess the overall response rate (ORR) of SG as well as compare the ORR of SG between homologous recombination-deficient (HRD) vs non-HRD in advanced TNBC patients, stratified by molecular subtypes using whole-genome and transcriptome analysis (WGTA). The 21-day cycle(s) treatment duration allows us to gather the necessary data to meet our primary and secondary objectives and exploratory endpoints. This study will be conducted in compliance with the protocol, the International Council of Harmonisation Good Clinical Practice guidelines, and every applicable regulatory requirement(s). This includes permitting study-related monitoring, audits, research ethics board review, and regulatory inspections, providing direct access to source data and documents.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible for participation in this study:

1. Willing and able to provide informed consent.
2. Age >18 years old at the time of informed consent and has signed informed consent before any trial related activities are conducted according to local guidelines.
3. For participants of child-bearing potential (menstruation within <2 years): negative serum pregnancy test within 14-days prior to enrollment and must be willing to use Health Canada-approved effective contraception methods (e.g., hormonal contraceptives, intrauterine device or system, tubal ligation, or double barrier method) starting 1 week prior to study treatment, throughout the study, and for 6 months following the last dose of SG.
4. For participants considered not of child-bearing potential (postmenopausal): must meet one of the following criteria at the time of study entry:

   i. Prior bilateral oophorectomy ii. Age > 60 iii. Age < 60 with >12 months of spontaneous amenorrhea (not due to chemotherapy, tamoxifen, toremifene, or ovarian suppression) and laboratory confirmation of postmenopausal FSH and estradiol levels per local postmenopausal reference ranges iv. Ovarian suppression with gonadotropin-releasing hormone (GnRH) agonist (e.g., goserelin) initiated >28 days before Cycle 1 Day 1
5. Advanced (locoregionally recurrent and non-operable, or metastatic) triple-negative breast cancer patients not amenable to curative therapy (surgery and/or radiotherapy), including those who are PDL1 negative (combined positive score [cps] <10), immuno-oncology therapy ineligible, or who had early-relapse after neoadjuvant therapy and not eligible for immuno-oncology in the first-line setting.
6. Histologically and/or cytologically confirmed diagnosis of estrogen-receptor negative breast cancer by local laboratory testing (based on most recently analyzed biopsy).
7. HER2-negative breast cancer (based on most recently analyzed biopsy) defined as negative in situ hybridization test or an immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, SISH) test is required by local laboratory testing, as defined in the relevant American Society of Clinical Oncology / College of American Pathologists Guidelines.
8. Not previously received systemic therapy in the advanced setting.
9. Participants can have measurable or non-measurable disease by CT or MRI as per RECIST Version 1.1 criteria as evaluated locally. Tumour lesions situated in a previously irradiated area are considered measurable if unequivocal progression has been documented in such lesions since radiation. All radiology studies must be performed within 28-days of Day 1 Cycle 1.
10. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
11. Life expectancy > 3 months.
12. Acceptable bone marrow and organ function defined by the following laboratory values without transfusion or growth factor support within 2 weeks of treatment initiation:

    a. Absolute neutrophil count > 1.0 x 109/L i. Platelets > 100 x 109/L ii. Hemoglobin > 90 g/dL iii. Potassium, sodium, calcium (corrected for serum albumin), and magnesium within normal limits.

    iv. INR < 1.5 v. Serum creatinine <1.5 x upper limit of normal (ULN) or calculated (Cockroft-Gault) or measured creatinine clearance ≥50 mL/min/1.73 m2 b. In absence of liver metastases, ALT and AST should be below <3.0 x ULN. If the participant has liver metastases, ALT and AST should be < 5.0 x ULN.

    c. In absence of liver metastases, total serum bilirubin < ULN; If the participant has liver metastases, total bilirubin < 3.0 x ULN with direct bilirubin < 1.5 x ULN.
13. Consents to allow access and provision of pre- and post-treatment biopsy specimens for study purposes.
14. Able to communicate with the Investigator and comply with the requirements of the study procedures.
15. Controlled brain metastasis (as per clinical determination) is allowed in the study at least 4 weeks before treatment. Controlled brain metastasis is defined as asymptomatic brain metastasis or no longer requiring high doses of corticosteroids (>10 mg Dexamethasone per day) for central nervous system (CNS) symptom management. Anticonvulsants and stable corticosteroids dose can be included in the study.

Waivers to the inclusion criteria will NOT be allowed.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Are within 4 weeks of participating in any other type of medical research judged by the Investigator to not be scientifically or medically compatible with this study.
2. Tumour not accessible or not safe to perform biopsies.
3. Has a known hypersensitivity to SG, irinotecan or its active metabolite SN-38.
4. Has received prior antibody-drug conjugate containing a topoisomerase 1 inhibitor.
5. Has a history of significant cardiovascular diseases, such as congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, serious cardiac arrhythmia, clinically significant electrocardiogram (ECG) findings or any other clinically significant cardiovascular condition, as determined by the Investigator.
6. Has a history or evidence of any condition or laboratory abnormality that would place the participant at undue risk, as determined by the Investigator.
7. Currently active Hepatitis B virus (HBV) or active Hepatitis C virus (HCV).

   1. For participants with a history of HBV infection, a hepatitis B core antibody test should be conducted at screening. If positive, hepatitis B DNA testing will be performed and if active HBV infection is ruled out, the participant may be eligible.
   2. Those who are HCV antibody positive with undetectable HCV viral load may be eligible.
8. Has an active human immunodeficiency virus (HIV) infection (e.g., with detectable viral load).

   a. Participants positive for HIV-1 or 2 with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
9. Has not had resolution of all acute toxic effects of prior anti-cancer therapy to CTCAE version 5.0 grade <1 (except toxicities not considered a safety risk for the participant at Investigator's discretion, e.g. grade 2 peripheral neuropathy from prior chemotherapy).
10. Have an active second malignancy. Participants with a history of malignancy that has been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or participants with surgically cured tumours with low risk of recurrence (e.g., non-melanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll.
11. Have known, untreated, active central nervous system (CNS) metastases. Participants with previously treated brain metastases may participate provided they have stable CNS disease, defined as no longer symptomatic from brain metastasis or no longer requires higher doses of corticosteroids (>10mg Dexamethasone per day) for CNS symptom management. Anticonvulsants and stable corticosteroids dose can be included in the study. Screening for brain metastasis is not required for enrollment.
12. Pregnancy or breast feeding.
13. Has inadequate hematologic, renal and hepatic function as outlined above in inclusion criteria.
14. Has a pre-existing condition with uncontrolled diarrhea, chronic inflammatory bowel disease (Ulcerative colitis, Crohn's Disease), or gastrointestinal perforation within 6-months prior to enrollment.
15. Has active serious infection requiring antibiotics.
16. Have other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may confound study interpretation or prevent completion of study procedures and follow-up examinations.
17. Received a live vaccine within 30 days prior to enrollment.
18. Current and/or prior use of systemic anticancer therapies, aside from the study drug. High-dose systemic corticosteroids (>20mg of prednisone or its equivalent) is not allowed within 2 weeks of Cycle 1 Day 1. Premedication with corticosteroids or the use of corticosteroids for treatment-related adverse events are permitted.
19. Persons of child-bearing potential (i.e., menstruation within < 2 years) who are unable or unwilling to use Health Canada approved highly effective methods of contraception (hormonal contraceptives, intrauterine device or system, vasectomy, tubal ligation, or double-barrier method), or abstinence during the treatment period and for 6 months following last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) of SG in advanced TNBC | Up to an average of 6 months
  To evaluate the overall response rate (ORR) of Sacituzumab govitecan (SG) in advanced triple-negative breast cancer (TNBC) patients without prior treatment in the advance setting, stratified by molecular subtypes using whole-genome and transcriptome analysis (WGTA).
ORR of SG between HRD vs non-HRD in advanced TNBC | Up to an average of 6 months
  2. To compare the ORR of SG between homologous recombination-deficient (HRD) vs non-HRD advanced TNBC patients without prior treatment in the advance setting, utilizing WGTA.

SECONDARY OUTCOMES:
Evaluate clinical benefit rate (CBR) of SG in advanced TNBC | Up to an average of 6 months
  To evaluate the clinical benefit rate (CBR) of SG in advanced TNBC, stratified by molecular subtypes identified through WGTA.
Assess progression-free survival (PFS) and overall-survival (OS) in advanced TNBC treated with SG | Up to an average of 12 months
  To assess progression-free survival (PFS) and overall survival (OS) in advanced TNBC patients receiving SG, stratified by molecular subtypes using WGTA.
Number of advanced TNBC participants receiving SG in first-line setting with treatment-related adverse events as assessed by CTCAE v5.0 | Up to an average of 3 months
  To assess the safety and toxicity profile in advanced TNBC participants receiving SG in the first-line setting per the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for grade 2-4 toxicities.
Changes in health-related quality of life when treated with SG | At follow-up, within 30 days following the last dose of study drug
  To assess changes in health-related quality of life using EORTC QLQ-CL30 version 3.0 questionnaire in advanced TNBC patients undergoing treatment with SG.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer - Vancouver Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldenberg DM, Sharkey RM. Antibody-drug conjugates targeting TROP-2 and incorporating SN-38: A case study of anti-TROP-2 sacituzumab govitecan. MAbs. 2019 Aug/Sep;11(6):987-995. doi: 10.1080/19420862.2019.1632115. Epub 2019 Jul 18. PMID 31208270
- [Background] Fenn KM, Kalinsky K. Sacituzumab govitecan: antibody-drug conjugate in triple-negative breast cancer and other solid tumors. Drugs Today (Barc). 2019 Sep;55(9):575-585. doi: 10.1358/dot.2019.55.9.3039669. PMID 31584574
- [Background] Bardia A, Hurvitz SA, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Sardesai SD, Kalinsky K, Zelnak AB, Weaver R, Traina T, Dalenc F, Aftimos P, Lynce F, Diab S, Cortes J, O'Shaughnessy J, Dieras V, Ferrario C, Schmid P, Carey LA, Gianni L, Piccart MJ, Loibl S, Goldenberg DM, Hong Q, Olivo MS, Itri LM, Rugo HS; ASCENT Clinical Trial Investigators. Sacituzumab Govitecan in Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2021 Apr 22;384(16):1529-1541. doi: 10.1056/NEJMoa2028485. PMID 33882206
- [Background] Sukumar J, Gast K, Quiroga D, Lustberg M, Williams N. Triple-negative breast cancer: promising prognostic biomarkers currently in development. Expert Rev Anticancer Ther. 2021 Feb;21(2):135-148. doi: 10.1080/14737140.2021.1840984. PMID 33198517
- See also: Sacituzumab govitecan (Trodelvy) Product Monograph — https://pdf.hres.ca/dpd_pm/00071772.PDF